CLINICAL TRIAL: NCT03111641
Title: Comparison of Lung Ultrasound Assessment and Chest Radiography During Perioperative Evaluation: a Prospective Study
Brief Title: The Role of Lung Ultrasound During Perioperative Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Francesco Forfori, Sponsor-Investigator, University of Pisa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPisa2017
Record Dates: First submitted 2017-04-02; First posted 2017-04-13 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung ultrasonography (Experimental)
  Interventions: Diagnostic Test: Lung ultrasonography

INTERVENTIONS:
Diagnostic Test: Lung ultrasonography — Lung ultrasound scan during preoperative anaesthesia consultation

SUMMARY:
Accurate pre-operative lung assessment is important to decide the most appropriate anesthesia plan. Until now, chest X-ray is considered the standard of care for lung assessment during perioperative evaluation. However, lung ultrasound is a rapid, simple, non-invasive, radiation-free imaging modality and can be used as an alternative to chest radiography for the diagnosis and follow-up of various lung diseases. Moreover, the decreased radiation exposure represents a considerable improvement in patient safety. Consequently, we decided to compare the data obtained from the lung ultrasound and the chest X-ray.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing elective general surgery;
* age >18 years;
* ability to provide written consent;
* use of Chest radiography during the preoperative evaluation.

Exclusion Criteria:

* age < than 18 year;
* pregnant patients;
* not use of Chest radiography during the preoperative evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-06-18 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Performance comparison of lung ultrasonography and chest x-ray in the detection of pleural effusion, consolidation, alveolar- interstitial syndrome. | during preoperative anaesthesia consultation
  The primary objective of this project is to evaluate the possible correlation between the data obtained from the ultrasound scan and the data obtained from the chest X-ray.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pisa, Pisa, Italy